CLINICAL TRIAL: NCT02399046
Title: A Prospective, Randomized, Multicenter, Controlled Study Comparing the Outcomes of Primary Total Knee Arthroplasty Devices Manufactured in China Versus Devices Manufactured Outside of China
Brief Title: A Clinical Trial Study of Knee System in Primary Total Knee Arthroplasty in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Medical (Suzhou) Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DPS-201302
Record Dates: First submitted 2015-03-20; First posted 2015-03-26 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Arthritis, Rheumatoid; Osteoarthritis; Post-traumatic; Arthrosis
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total Knee System made in China (Experimental): Patinet in this arm will be implanted with Primary Total Knee Arthroplasty Devices Manufactured in China
  Interventions: Device: Total Knee System made in China (Sigama, CoCr, PFC)
- Total Knee System made outside of China (Active Comparator): Patient in this arm will be implanted with Primary Total Knee Arthroplasty Devices Manufactured Outside of China
  Interventions: Device: Total Knee System made outside of China (Sigama, NP, PFC)

INTERVENTIONS:
Device: Total Knee System made in China (Sigama, CoCr, PFC) — SIGAMA PS FEMUR; TIB tray Cem Cocr; SIGAMA STAB XLK INS; PFC SIG ROUND DOME PAT 3PEG
  Arms: Total Knee System made in China
Device: Total Knee System made outside of China (Sigama, NP, PFC) — SIGAMA PS CEM FEM; PFC MOD TIB TRAY NP; SIGAMA STAB XLK INS; PFC SIGAMA/RD/DOME PAT
  Arms: Total Knee System made outside of China

SUMMARY:
A clinical trial of total knee system used in Primary Total Knee Arthroplasty in China.

DETAILED DESCRIPTION:
A prospective, Randomized, Multicenter, Controlled Study Comparing the Outcomes of Primary Total Knee Arthroplasty Devices Manufactured in China versus Devices Manufactured Outside of China.

ELIGIBILITY:
Inclusion Criteria:

1. . The subject is ≥18years old
2. . The Subject must be of Chinese ethnic descent and be willing to return on three occasions for clinical evaluations.
3. . Subject is a suitable candidate for cemented primary TKA using the devices described in this CIP with either resurfaced or non-resurfaced patellae.
4. . Subject must meet all criteria specified in BOTH China Knee stem and P.F.C.® Sigma knee instructions for use (IFU)
5. . Before surgery, subject is willing and able to sign the informed consent form approved by the Institutional Review Board (IRB), Ethics Committee (EC) or Ethical Review Board (ERB).
6. . Subject, in the opinion of the Clinical Investigator, is able to understand this clinical investigation and co-operate with investigational procedures.
7. . Subject must be comfortable with speaking, reading, and understanding questions and providing responses in an available translated language for the patient reported outcomes (PROs) in the CIP.
8. . Subject is receiving a unilateral knee replacement or, if a contralateral knee replacement is anticipated, the surgery must occur within 6 months of the first study knee TKA. The second knee will not be enrolled in the study.

Exclusion Criteria:

1. Subject does not provide written voluntary consent to participate in the clinical study.
2. The Subject is a woman who is pregnant or lactating.
3. Subject is anticipated to require a contralateral TKA between 6 months and 1 year.
4. Contralateral knee has already been enrolled in this study.
5. Previous partial knee replacement (unicompartmental, bicompartmental or patellofemoral joint replacement), patellectomy, high tibial osteotomy or primary TKA in affected knee.
6. Subject has a malignant disease, severe condition, alcohol or drug addiction and/or mental disorders that the investigator believes will interfere with the study participation.
7. Subjects with severe osteoporosis, metabolic bone disease, radioactive bone disease or tumor in bone surrounding knee joint that, in the opinion of the investigator, will negatively impact implant fixation and the outcome of the investigation
8. Subject has significant neurological or musculoskeletal disorders or disease that may adversely affect gait or weight bearing (e.g. muscular dystrophy, multiple sclerosis, cerebral infarction, hemiplegia, Charcot disease).
9. Subject is not comfortable with speaking, reading, and understanding questions and providing responses in an available translated language for the PROs in the CIP.
10. Subject has a medical condition with less than 2 years of life expectancy.
11. The Subject has comorbid condition(s) that could limit the Subject's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study.
12. The Subject is currently participating in another investigational drug or device study.
13. Subject is a prisoner.
14. The Subject has a known allergy to any implant components (metal for example).
15. Hemoglobin < 11 g/dL
16. Albumin < 90% normal low limit
17. CRP > 2 times normal upper limit
18. ESR > 2 times normal upper limit
19. Subjects who have abnormal coagulation exam results and cannot be corrected by drugs or plasma replacement

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
12-month post-op AKS | 12 months postoperatively

SECONDARY OUTCOMES:
Non-revision rates(revision for any reason) through the end of the study | 12 months postoperatively
One year non-revision rate where revision is defined as removal of any component secondary to infection | 12 months postoperatively
American Knee Society Total Score success (where success is defined as a score of 80 points or higher)at the 1 year follow-up inerval | 12 months postoperatively
Short-form 12(SF-12) general health questionnaire each of 8 dimensions and the overall Physical and Mental health domains, at 1-year follow-up interval. | Preoperation to12 months postoperatively
WOMAC scores at the 1-year follow-up interval | Preoperation to12 months postoperatively
Radiogrphic assessment of clinically relevant radiolucent line(RLL)and osteolysis,migration and subsidence, by comparing the 3 month post-operative x-ray to the 1 year follow up x-ray inerval. | Preoperation to12 months postoperatively

OTHER OUTCOMES:
The proportion of Composite Successes in each treatment group will be assessed at the 1year follow-up interval | 12 months postoperatively
Blood samplets will be collected and data will be summarized | pre-operative and immediate post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Fuxing Pei, Principal Investigator — The West China Hospital of Sichuan University
Locations (9):
- China (9):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - General Hospital of Guangzhou Military Command of PLA, Guangzhou, Guangdong
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The affiliated hosoital of Ningxia Medical University, Yinchuan, Ningxia
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Xijing Hospital, Xi’an, Shanxi
  - The West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang